CLINICAL TRIAL: NCT06820918
Title: Impact of Physiotherapy With Positive Expiratory Pressure (PEP) Bottle on Respiratory Function in Patients With Bronchiectasis (FisioFEV)
Brief Title: Physiotherapy With Positive Expiratory Pressure (PEP) Bottle in Patients With Bronchiectasis
Acronym: FisioFEV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6836
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with bronchiectasis (Experimental)
  Interventions: Device: Bottle PEP

INTERVENTIONS:
Device: Bottle PEP — Home respiratory physiotherapy using the PEP bottle for a minimum of 10 minutes to a maximum of 30 minutes, twice a day (morning and evening), every day for 30 days

SUMMARY:
The aim of this study is to determine whether respiratory physiotherapy using the Positive Expiratory Pressure (PEP) bottle has an effect on respiratory function, measured through spirometry, in patients with a diagnosis of bronchiectasis not associated with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Confirmed diagnosis of bronchiectasis based on high-resolution chest CT, showing bronchial dilation according to one or more of the following radiological criteria in accordance with the 2019 BTS guidelines.
* Ratio between the internal lumen of the bronchus and the adjacent pulmonary artery >1
* Absence of normal bronchial tapering
* Visibility of the airways within 1 cm from the pleura
* Subject with chronic bronchial hypersecretion (daily secretion ≥ 15ml)
* Patients capable of performing physiotherapy using the PEP bottle
* Patients capable of performing global spirometry

Exclusion Criteria:

* Subject already undergoing regular respiratory physiotherapy
* Subject without significant bronchial hypersecretion
* Concomitant diagnosis of Cystic Fibrosis, Primary Ciliary Dyskinesia, NTM-PD, TB, Sarcoidosis, Active Neoplasia
* Diagnosis of Asthma according to the 2023 GINA guidelines, defined as documented excessive variability in pulmonary function (positive bronchodilation or bronchoprovocation test with methacholine, or diurnal variability of PEF) + documented limitation of expiratory airflow.
* Diagnosis of COPD according to the 2023 GOLD guidelines, defined as FEV/FVC post-bronchodilation <0.7 on forced spirometry in the presence of suggestive symptoms (dyspnea, chronic cough, sputum production) and/or exposure to risk factors for the disease (e.g., cigarette smoking).
* Contraindications to PEP-Bottle Physiotherapy (Pneumothorax; Hemoptysis; Myocardial infarction in the 4 weeks prior to informed consent signature)
* Exacerbation of disease in the previous 4 weeks
* Use of inhalation therapy in the 4 weeks prior to informed consent signature
* Active smoker
* Subject undergoing non-invasive ventilation or with a tracheostomy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of respiratory physiotherapy using a PEP bottle on respiratory function through the measurement of FEV1 (Forced Expiratory Volume in the 1st second) | 60 days
  To evaluate the effect of respiratory physiotherapy using the PEP bottle on respiratory function in patients with a diagnosis of bronchiectasis not associated with cystic fibrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy